CLINICAL TRIAL: NCT00583986
Title: A Study to Determine the Reliability of a Top Mount Actuation Indicator When Used With Levalbuterol Tartrate HFA MDI in Adult and Pediatric Subjects With Asthma or Chronic Obstructive Pulmonary Disease
Brief Title: Reliability of a Top Mount Actuation Indicator With Levalbuterol MDI in Adult and Pediatric Subjects With Asthma or COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 051-357
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease; COPD
Keywords: top mounted; actuation indicator; Asthma; COPD; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Levalbuterol HFA MDI with top mounted actuation indicator
  Interventions: Drug: Levalbuterol HFA MDI with top mounted actuation indicator

INTERVENTIONS:
Drug: Levalbuterol HFA MDI with top mounted actuation indicator — Levalbuterol HFA MDA with top mounted actuation indicator
  Other Names: Xopenex HFA®

SUMMARY:
This is a study to investigate the reliability, ruggedness and safety of the top mounted actuation indicator (TMAI) when used with Levalbuterol HFA MDI.

DETAILED DESCRIPTION:
This is an open-label, multicenter, TMAI study with Levalbuterol HFA MDI in adult and pediatric subjects with asthma or COPD. Period I: One week, open-label, run-in period during which subjects must have asthma or COPD symptoms requiring use of, as needed, Levalbuterol HFA MDI(without TMAI) on at least half of the days [4-12 actuations on a single day]. Period II: Nine week, open-label period during which subjects will use the Levalbuterol HFA MDI with TMAI PRN. The total study duration for a subject will not exceed 10 weeks. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a documented diagnosis of asthma or COPD for a minimum of 6 months.
* Subject must have stable baseline asthma or COPD and have been using a beta-adrenergic agonist, and/or anti-asthma anti-inflammatory medication, and/or over-the-counter asthma medication for at least 6 months.
* Subject must be in good health with the exception of their reversible airways disease and not suffering from any chronic condition that might affect their respiratory function.

Exclusion Criteria:

* Female subject who is pregnant or lactating.
* Subject who has a history of hospitalization for asthma or COPD within 45 days.
* Subject with currently diagnosed life-threatening asthma or COPD, defined as a history of asthma or COPD episodes requiring intubation, associated with hypercapnia, respiratory arrest, or hypoxic seizures within 3 months prior.
* Subject with supplemental oxygen use
* Subject with a history of cancer
* Subject with hyperthyroidism, diabetes, hypertension, cardiac diseases, or seizure disorders that currently are not well controlled by medication.
* Subject with asthma with a greater than 10-pack per year history of cigarette smoking or use of any tobacco products within 6 months.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-09; Primary Completion 2006-01 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The difference between the number of actuations estimated via canister weight and the number of actuations recorded byt eh TMAI. | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Hanrahan, M.D., Study Chair — Sumitomo Pharma America, Inc.
Locations (26):
- United States (26):
  - Encinatas, California
  - Huntington Beach, California
  - Mesa, California
  - Orange County, California
  - Riverside, California
  - San Diego, California
  - San Jose, California
  - Viejo, California
  - Walnut Creek, California
  - Tamarac, Florida
  - Russells Mills, Massachusetts
  - Commack, New York
  - Rochester, New York
  - Elizabeth City, North Carolina
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Simpsonville, South Carolina
  - Chattanooga, Tennessee
  - Austin, Texas
  - Braunfels, Texas
  - San Antonio, Texas
  - Burke, Virginia
  - Richmond, Virginia
  - Morgantown, West Virginia

REFERENCES:
- See also: Patient's Instructions for Use — http://www.xopenex.com/about/patient-instructions.html